CLINICAL TRIAL: NCT03347175
Title: Pilot Study: Comparison of Ventilation Modes During Cardio-pulmonary Resuscitation With a Mechanical Compression Device in the Emergency Room
Brief Title: Pilot Study Comparing Ventilation Modes During CPR With Mechanical Compression Device.
Acronym: COVME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Stefan Schaller, Principal Investigator, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVME
Record Dates: First submitted 2017-10-24; First posted 2017-11-20 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: Respiration, Artificial; Advanced Cardiac Life Support; Heart Massage; Emergency Service, Hospital
MeSH Terms: conditions — Respiratory Aspiration; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Volume controlled ventilation (Experimental): Intervention1: Ventilation with Volume controlled ventilation
  Interventions: Procedure: Volume controlled ventilation
- Pressure controlled ventilation (Active Comparator): Intervention2: Ventilation with Pressure controlled ventilation
  Interventions: Procedure: Pressure controlled ventilation
- CPAP mode (Active Comparator): Intervention3: Ventilation with Continuous Positive Airway Pressure mode only
  Interventions: Procedure: CPAP mode

INTERVENTIONS:
Procedure: Volume controlled ventilation — Volume controlled ventilation mode
  Arms: Volume controlled ventilation
Procedure: Pressure controlled ventilation — Pressure controlled ventilation
  Arms: Pressure controlled ventilation
Procedure: CPAP mode — CPAP mode only
  Arms: CPAP mode

SUMMARY:
Comparison of three ventilation modes (volume controlled, BIPAP and CPAP) during cardiopulmonary re-suscitation with a mechanical compression device in the emergency room. Primary aim is to assess mean ventilation volume in the first 15 minutes after randomization.

DETAILED DESCRIPTION:
Mechanical compression devices are applied to grant continuous chest compressions and consequently blood flow during CPR (cardiopulmonary rescuscitation). Current guidelines, however, are lacking guidance of the optimal ventilation strategy in such scenarios. This may lead to lung injuries caused by high pressure levels in the chest while applying compression and ventilation simultaneously or hypoventilation. Consequently, this pilot study assesses iwhich ventilation mode is optimal. Patients will be assigned randomly to one of the three ventilation modes (Volume controlled, BiPAP-ASB, CPAP). Ventilation parameters will be continuously monitored for 15 minutes while blood gas analyses are taken as well. Further secondary outcome parameters will be assessed, e.g. hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* On-going out of hospital CPR in the Emergency Room
* Tracheal intubated
* Use of mechanical chest compression device

Exclusion Criteria:

* If the treating team assumes that CPR will be ceased within the next 15 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
mean tidal volume | Study period = 15 min (Startpoint = Activating randomized ventilation mode Endpoint = 15 minutes after Starting point or end of CPR)
  mean tidal volume during the study period

SECONDARY OUTCOMES:
mean minute volume | Study period = 15 min (Startpoint = Activating randomized ventilation mode Endpoint = 15 minutes after Starting point or end of CPR)
  mean minute volume during the study period
etCO2 | Study period = 15 min (Startpoint = Activating randomized ventilation mode Endpoint = 15 minutes after Starting point or end of CPR)
  Mean, final value and course of the parameter during the study period

OTHER OUTCOMES:
paO2 | Study period = 15 min (Startpoint = Activating randomized ventilation mode Endpoint = 15 minutes after Starting point or end of CPR)
  Mean, final value and course of the parameter during the study period
paCO2 | Study period = 15 min (Startpoint = Activating randomized ventilation mode Endpoint = 15 minutes after Starting point or end of CPR)
  Mean, final value and course of the parameter during the study period
Ventilation setting change | Study period = 15 min (Startpoint = Activating randomized ventilation mode Endpoint = 15 minutes after Starting point or end of CPR)
  We will assess changes made in the ventilator settings (mode, tidal volume, frequency, FiO2 and PEEP) during the study period
Ventilation setting change lateron | Starting after the end of Study Period (15 min after randomized ventilation mode was activated) till cardiopulmonary resuscitation is stopped by the treating team
  We will assess changes made in the ventilator settings (mode, tidal volume, frequency, FiO2 and PEEP) after study period until the end of CPR
Ventilation hours | Starting point = Activation of randomized ventilation mode till End point = time when patient is discharged from the hospital; ; approximately 3 weeks
  Ventilation hours in the hospital
24h Survival | 24h after randomization
  Survival 24h after randomization
Hospital Survival/Mortality | Starting point = Activation of randomized ventilation mode till End point = time when patient is discharged from the hospital; approximately 3 weeks
  Hospital Survival/Mortality
BGA | Study period = 15 min (Startpoint = Activating randomized ventilation mode Endpoint = 15 minutes after Starting point or end of CPR)
  Blood gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Klinik für Anaesthesiologie
Locations (1):
- Klinikum rechts der Isar, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
We are willing to share anonymized and aggregated data for meta analysis or on an individual decision to collaboration partners.

REFERENCES:
- [Background] Bernhard M, Hossfeld B, Kumle B, Becker TK, Bottiger B, Birkholz T. Don't forget to ventilate during cardiopulmonary resuscitation with mechanical chest compression devices. Eur J Anaesthesiol. 2016 Aug;33(8):553-6. doi: 10.1097/EJA.0000000000000426. No abstract available. PMID 26854661
- [Background] Hillman K, Albin M. Pulmonary barotrauma during cardiopulmonary resuscitation. Crit Care Med. 1986 Jul;14(7):606-9. doi: 10.1097/00003246-198607000-00003. PMID 3720308
- [Background] Shulman D, Beilin B, Olshwang D. Pulmonary barotrauma during cardiopulmonary resuscitation. Resuscitation. 1987 Sep;15(3):201-7. doi: 10.1016/0300-9572(87)90015-3. PMID 2823358
- [Background] Hou SH, Lue HC, Chu SH. Comparison of conventional and simultaneous compression-ventilation cardiopulmonary resuscitation in piglets. Jpn Circ J. 1994 Jun;58(6):426-32. doi: 10.1253/jcj.58.426. PMID 8065014
- [Background] Kleinsasser A, Lindner KH, Schaefer A, Loeckinger A. Decompression-triggered positive-pressure ventilation during cardiopulmonary resuscitation improves pulmonary gas exchange and oxygen uptake. Circulation. 2002 Jul 16;106(3):373-8. doi: 10.1161/01.cir.0000021428.94652.04. PMID 12119256
- [Background] Kill C, Hahn O, Dietz F, Neuhaus C, Schwarz S, Mahling R, Wallot P, Jerrentrup A, Steinfeldt T, Wulf H, Dersch W. Mechanical ventilation during cardiopulmonary resuscitation with intermittent positive-pressure ventilation, bilevel ventilation, or chest compression synchronized ventilation in a pig model. Crit Care Med. 2014 Feb;42(2):e89-95. doi: 10.1097/CCM.0b013e3182a63fa0. PMID 24158168
- [Background] Winkler BE, Muellenbach RM, Wurmb T, Struck MF, Roewer N, Kranke P. Passive continuous positive airway pressure ventilation during cardiopulmonary resuscitation: a randomized cross-over manikin simulation study. J Clin Monit Comput. 2017 Feb;31(1):93-101. doi: 10.1007/s10877-016-9836-6. Epub 2016 Feb 9. PMID 26861639
- [Background] Kill C, Galbas M, Neuhaus C, Hahn O, Wallot P, Kesper K, Wulf H, Dersch W. Chest Compression Synchronized Ventilation versus Intermitted Positive Pressure Ventilation during Cardiopulmonary Resuscitation in a Pig Model. PLoS One. 2015 May 26;10(5):e0127759. doi: 10.1371/journal.pone.0127759. eCollection 2015. PMID 26011525
- [Background] Tan D, Xu J, Shao S, Fu Y, Sun F, Zhang Y, Hu Y, Walline J, Zhu H, Yu X. Comparison of different inspiratory triggering settings in automated ventilators during cardiopulmonary resuscitation in a porcine model. PLoS One. 2017 Feb 10;12(2):e0171869. doi: 10.1371/journal.pone.0171869. eCollection 2017. PMID 28187154